CLINICAL TRIAL: NCT06319157
Title: A Randomized Controlled Study of Minimal Access Latissimus Dorsi Flap Harvest for Breast Reconstruction Versus Conventional Approaches in the Treatment of Early Breast Cancer
Brief Title: Minimal Access Versus Conventional Latissimus Dorsi Flap Harvest for Breast Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-1263-02
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- minimal access group (Experimental)
  Interventions: Device: minimal access breast reconstruction with a latissimus dorsi muscle flap
- conventional group (Other)
  Interventions: Device: conventional breast reconstruction with a latissimus dorsi muscle flap

INTERVENTIONS:
Device: minimal access breast reconstruction with a latissimus dorsi muscle flap — minimal access breast reconstruction with a latissimus dorsi muscle flap
  Arms: minimal access group
Device: conventional breast reconstruction with a latissimus dorsi muscle flap — conventional breast reconstruction with a latissimus dorsi muscle flap
  Arms: conventional group

SUMMARY:
For patients refusing implants for breast reconstruction after cancer surgery, autologous tissue flap reconstruction using the latissimus dorsi muscle is an alternative. Conventional surgery leaves a long incision on the back, affecting aesthetics and quality of life. Minimal access techniques result in a smaller, more concealable scar. While previous studies suggest its safety and effectiveness, most are retrospective. To further validate patient satisfaction and short-term outcomes, a prospective, randomized controlled trial comparing minimal access with conventional surgery is planned. The primary endpoint is Breast Q-satisfaction with back score at 6 months. Secondary outcomes include other Breast Q subscales, surgical metrics, and complications. The study aims to enroll 94 patients in total, providing evidence for surgical decision-making in breast cancer reconstruction.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with early-stage breast cancer between the ages of 18 and 70.
2. Breast cancer was confirmed by histology or biopsy.
3. Breast-conserving surgery or multifocal breast cancer or large unifocal breast cancer (<5cm) can be accepted.
4. After neoadjuvant therapy, large monofocal carcinoma (>5 cm) confined to the breast shrunk to <5 cm.
5. No chest wall, cutaneous or NAC invasion (including Paget's disease).
6. Mild to moderate breast sagging, and the patient has the willingness to undergo autologous reconstruction of the latissimus dorsi.
7. There is no need to obtain additional back skins.
8. Willing to participate and able to complete follow-up and evaluation during the study.

Exclusion Criteria:

1. Patients with advanced breast cancer (stage III and above) or metastatic breast cancer or inflammatory breast cancer.
2. The risk of recurrence is expected to be high.
3. History of thoracic and dorsal vascular injury.
4. Patients with severe heart, lung, or liver disease who cannot withstand surgery and anesthesia.
5. Patients with active infection or severe immune system disease.
6. Patients with severe allergic reactions to materials related to latissimus dorsi muscle flap transplantation.
7. Patients with other major surgeries or reconstructive surgeries planned for the near future.
8. Patients with cognitive dysfunction or psychiatric disorders who cannot understand and cooperate with the requirements of the study.
9. Patients who refuse to participate in the study or are unable to complete follow-up and evaluation during the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Breast Q-satisfaction with back | 6 months
  Patient satisfaction with the back, assessed using the Breast Q-satisfaction with back subscale.
  6 months after surgery, the doctor provided each patient with a Breast Q-satisfaction with back questionnaire, and asked the patient to fill in the questionnaire truthfully, and each questionnaire took 1-4 minutes to complete. Before each questionnaire is completed, the doctor will give the patient a simple guide to make it clear what each option means.

SECONDARY OUTCOMES:
Patient satisfaction | 6 months
  Other aspects of patient satisfaction, assessed using the Breast Q scale. 6 months after surgery, the doctor provided each patient with a questionnaire and asked the patient to fill it out truthfully, each questionnaire takes 1-4 minutes to complete, and a complete BREAST-Q survey can be completed in 10-15 minutes. Before each questionnaire is completed, the doctor will give the patient a simple guide to make it clear what each option means.
Latissimus dorsi acquisition time | Perioperative
  Calculated from the start of latissimus dorsi acquisition to the completion of latissimus dorsi acquisition.
Intraoperative blood loss | Perioperative
  The amount of blood lost by the patient due to routine operations during surgery.
Postoperative pain | Perioperative
  recorded using the Visual Analogue Scale (VAS) pain assessment tool.
Postoperative complications | 6 months
  including but not limited to surgical site infection, bleeding, wound dehiscence, breast/donor site flap/NAC necrosis, subcutaneous effusion in the chest and donor site, surgical side lymphedema, etc., are classified using the Clavien-Dindo grading system.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China